CLINICAL TRIAL: NCT02237911
Title: A Comparison of Treatment Methods for Patients Following Total Knee Replacement.
Brief Title: Comparison of Treatments Following Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Sara R. Piva, Dr., University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO14080261; CER-1310-06994 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2018-11

CONDITIONS: Degeneration; Articular Cartilage, Knee; Rheumatoid Arthritis; Osteoarthritis, Knee
Keywords: total knee replacement; rehabilitation; exercise program; total knee arthroplasty
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Clinic-based outpatient exercise group (Experimental): Subjects will participate in supervised sessions (clinic-based) of exercise followed by a home exercise program 2 times per week during 3 months. Each exercise session will last about 60 minutes. Treatment sessions will utilize a pragmatic approach and will include the exercises designed to increase muscular strength, low impact cardiovascular exercise, range of movement, and activity for daily living skills.
  Interventions: Other: Clinic-based outpatient exercise group
- Community-based exercise group (Active Comparator): Subjects will attend to exercise classes (community-based) 2 times per week during 3 months. The exercise classes last approximately 60 minutes. The group exercise classes consists of a variety of exercises designed to increase general muscular strength, low impact aerobic exercise, range of movement, and activity for daily living.
  Interventions: Other: Community-based exercise group
- Wait-listed usual medical care (No Intervention): Wait-listed usual medical care - no intervention provided by study.

INTERVENTIONS:
Other: Clinic-based outpatient exercise group — Subjects will participate in supervised sessions (clinic-based) of exercise followed by a home exercise program 2 times per week during 3 months. Each exercise session will last about 60 minutes. Treatment sessions will utilize a pragmatic approach and will include the exercises designed to increase muscular strength, low impact cardiovascular exercise, range of movement, and activity for daily living skills.
  Arms: Clinic-based outpatient exercise group
Other: Community-based exercise group — Subjects will attend to exercise classes (community-based) 2 times per week during 3 months. The exercise classes last approximately 60 minutes. The group exercise classes consists of a variety of exercises designed to increase general muscular strength, low impact aerobic exercise, range of movement, and activity for daily living.
  Arms: Community-based exercise group

SUMMARY:
Although total knee replacement (TKR) improves pain in numerous patients, it does not resolve many of the substantial functional limitations and physical inactivity that existed for a long time prior to the surgery. Exercise is an intervention that could improve these long-term limitations. To promote these improvements, exercise should be implemented at later stage post TKR when patients can tolerate doses of exercise sufficiently high to promote substantial changes. To date, we just don't have enough good research to tell us which type of exercise works best for which patients and under which circumstances at later stage post TKR. This research study will provide evidence for recommended interventions during the later stage post TKR. The specific research questions are: (1) How do group exercise in the community and individual exercise in rehabilitation clinic compare with usual medical care on physical function and activity outcomes? (2) Who are the patients most likely to respond to each exercise intervention? (3) Are the approaches safe?

DETAILED DESCRIPTION:
This is a comparative effectiveness study, designed as a 3-group single-blind randomized clinical trial. Two hundred forty older adults who underwent TKR at least 2 months prior and are otherwise eligible will be randomized into one of three treatment approaches: 1) clinic-based individual outpatient rehabilitative exercise; 2) community-based group exercise classes; or 3) usual medical care. Subjects will be treated for 3 months. Data will be collected before intervention, after intervention (3 months), and 6 months after randomization. Physical function is a primary outcome and will be assessed by the Western Ontario and McMaster Universities Arthritis Index and a battery of performance-based tests germane to patients post TKR that includes ability to walk, manage stairs, lift from the floor and the chair, and one-leg balance. We will also use an accelerometer-based monitor that provides a real-time measure of physical activity during normal daily living and is able to accurately capture most levels of activity. Linear mixed models will be fitted to compare the changes in outcome across groups. Logistic regression will identify patient characteristics that predict functional recovery in the exercise groups. Survival analysis and instrumental variable methods will be used to compare attrition, adherence and adverse events between groups.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral TKR 2 to 4 months prior
* Older than 60 years of age
* Experience functional limitation in daily activities (score in WOMAC-PF of at least 9 points)
* Speak sufficient English to understand study instructions
* Have medical clearance to participate in the study
* Are willing to be randomized to one of the 3 treatment arms

Exclusion Criteria:

* Have absolute or relative contraindications to exercise
* Have history of uncontrolled cardiovascular disease or hypertension
* Are unable to walk 50 meters without an assistive device
* Have history of muscular or neurological disorder that affect lower extremity function
* Regular participation in exercise
* Terminal illness
* Planning to have another joint replacement during the next 12 months
* Plan not to be around during the next 12 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2014-12; Primary Completion 2017-09-07 (Actual); Study Completion 2017-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara R Piva, PT, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Department of Physical Therapy, University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Piva SR, Schneider MJ, Moore CG, Catelani MB, Gil AB, Klatt BA, DiGioia AM, Almeida GJ, Khoja SS, Sowa G, Irrgang JJ. Effectiveness of Later-Stage Exercise Programs vs Usual Medical Care on Physical Function and Activity After Total Knee Replacement: A Randomized Clinical Trial. JAMA Netw Open. 2019 Feb 1;2(2):e190018. doi: 10.1001/jamanetworkopen.2019.0018. PMID 30794296
- [Derived] Piva SR, Moore CG, Schneider M, Gil AB, Almeida GJ, Irrgang JJ. A randomized trial to compare exercise treatment methods for patients after total knee replacement: protocol paper. BMC Musculoskelet Disord. 2015 Oct 16;16:303. doi: 10.1186/s12891-015-0761-5. PMID 26474988

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential subjects were identified from their surgeons' office or via public announcement in the greater Pittsburgh area, from December 2014 through February 2017. If interested in the study, subjects called the research team to obtain more information about the study, and were then screened for study eligibility.
Pre-assignment Details: A total of 1372 subjects called for study information: 89 could not be contacted and 1283 were screened over the telephone. From those, 1032 were not eligible/willing to participate and 251 completed in-person screening. Eleven subjects failed in-person screening, resulting in 240 eligible subjects that were randomized into one of the study arms.
Groups:
- Clinic-based Outpatient Exercise Group: Subjects participated in supervised sessions (clinic-based) of exercise followed by a home exercise program 2 times per week during 3 months. Each exercise session lasted about 60 minutes. Treatment sessions utilized a pragmatic approach and included the exercises designed to increase muscular strength, low impact cardiovascular exercise, range of movement, and activity for daily living skills.
- Community-based Exercise Group: Subjects attended to exercise classes (community-based) 2 times per week during 3 months. The exercise classes lasted approximately 60 minutes. The group exercise classes consisted of a variety of exercises designed to increase general muscular strength, low impact aerobic exercise, range of movement, and activity for daily living.
Period: Overall Study
Arm/Group | Clinic-based Outpatient Exercise Group | Community-based Exercise Group | Wait-listed Usual Medical Care
Started | 96 | 96 | 48
3 Months | 90 | 87 | 44
6 Months | 89 | 88 | 45
Completed | 89 | 88 | 45
Not Completed | 7 | 8 | 3
Not completed — Withdrawal by Subject | 4 | 7 | 2
Not completed — Lost to Follow-up | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Clinic-based Outpatient Exercise Group: Subjects participated in supervised sessions (clinic-based) of exercise followed by a home exercise program 2 times per week during 3 months. Each exercise session lasted about 60 minutes. Treatment sessions utilized a pragmatic approach and included exercises designed to increase muscular strength, low impact cardiovascular exercise, range of movement, and activity for daily living skills.
- Total: Total of all reporting groups
Arm/Group | Clinic-based Outpatient Exercise Group | Community-based Exercise Group | Wait-listed Usual Medical Care | Total
Number analyzed (Participants) | 96 | 96 | 48 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (6.3) | 70 (7.0) | 70 (6.6) | 70 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 58 | 31 | 148
  Male | 37 | 38 | 17 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 96 | 95 | 47 | 238
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 18 | 11 | 39
  White | 86 | 77 | 37 | 200
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Education [Count of Participants; unit: Participants]
  Less than college | 31 | 33 | 12 | 76
  Complete college or technical training | 59 | 57 | 31 | 147
  Other/missing | 6 | 6 | 5 | 17
Marital status [Count of Participants; unit: Participants]
  Married | 64 | 62 | 31 | 157
  Divorced | 18 | 12 | 7 | 37
  Widowed | 8 | 14 | 6 | 28
  Never Married | 4 | 8 | 3 | 15
  Other | 2 | 0 | 1 | 3
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.8 (5.3) | 31.1 (6.3) | 31.5 (5.1) | 31.1 (5.7)
Cumulative Illness Rating Scale [Mean (Standard Deviation); unit: Number of comorbidities] | 4.3 (2.0) | 4.4 (1.7) | 4.6 (1.9) | 4.4 (1.9)
Total Knee Replacement Due To [Count of Participants; unit: Participants]
  Osteoarthritis | 92 | 92 | 48 | 232
  Inflammatory Arthritis | 4 | 4 | 0 | 8
Surgical Knee Flexion [Mean (Standard Deviation); unit: degrees] | 124 (11) | 123 (11) | 124 (10) | 124 (11)
Surgical knee pain [Mean (Standard Deviation); unit: units on a scale] — Numeric Pain Rating Scale (NPRS). Current pain intensity was measure by NRPS. Score ranged from 0 to 10, 0 representing no pain, and 10 representing worse pain imaginable.
  units on a scale | 2.7 (2.1) | 2.3 (1.7) | 2.2 (1.8) | 2.4 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: The Western Ontario and McMaster Universities Osteoarthritis Index Physical Function (WOMAC-PF).
Description: WOMAC-PF is a patient reported outcome with 17 items. Each item is scored on a 5-point Likert-type Scale with descriptors from 0-4 (none, mild, moderate, severe, and extreme difficulty) and summed for a maximum score of 68. Higher scores indicate worse physical function.
Time Frame: Baseline, 3 and 6 months
Population: Intention-to-treat approach was used among participants with follow-up data.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Clinic-based Outpatient Exercise Group: Clinic-based outpatient exercise group: Subjects participated in supervised sessions (clinic-based) of exercise followed by a home exercise program 2 times per week during 3 months. Each exercise session lasted about 60 minutes. Treatment sessions utilized a pragmatic approach and will include the exercises designed to increase muscular strength, low impact cardiovascular exercise, range of movement, and activity for daily living skills.
- Community-based Exercise Group: Community-based exercise group: Subjects attended to exercise classes (community-based) 2 times per week during 3 months. The exercise classes lasted approximately 60 minutes. The group exercise classes consists of a variety of exercises designed to increase general muscular strength, low impact aerobic exercise, range of movement, and activity for daily living.
Arm/Group | Clinic-based Outpatient Exercise Group | Community-based Exercise Group | Wait-listed Usual Medical Care
Number analyzed (Participants) | 96 | 96 | 48
units on a scale
  Baseline | 20.9 (7.9) | 20.4 (7.4) | 20.2 (7.9)
  3 months: number analyzed (Participants) | 90 | 87 | 44
  3 months | 10.1 (6.6) | 12.2 (7.9) | 11.9 (7.6)
  6 months: number analyzed (Participants) | 89 | 88 | 45
  6 months | 9.8 (7.2) | 10.8 (7.9) | 11.8 (7.5)
Statistical Analysis 1: Comparison: Clinic-based Outpatient Exercise Group vs Wait-listed Usual Medical Care; Test type: Superiority; p = 0.071, Mixed Models Analysis; Contrasts from a linear mixed models analysis at 3 months adjusted for randomization factors (age, gender, BMI, WOMAC-PF, knee flexion); Mean Difference (Final Values) = -2.1, 98.3% CI 2-sided [-4.9 to 0.7]
Statistical Analysis 2: Comparison: Clinic-based Outpatient Exercise Group vs Wait-listed Usual Medical Care; Contrasts from a linear mixed models analysis at 6 months adjusted by baseline age, gender, BMI, WOMAC-PF, knee flexion; Test type: Superiority; p = 0.074, Mixed Models Analysis; Mean Difference (Final Values) = -2.1, 98.3% CI 2-sided [-5.0 to 0.7]
Statistical Analysis 3: Comparison: Community-based Exercise Group vs Wait-listed Usual Medical Care; Contrasts from a linear mixed models analysis at 3 months adjusted by baseline age, gender, BMI, WOMAC-PF, knee flexion; Test type: Superiority; p = 0.930, Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 98.3% CI 2-sided [-2.7 to 2.9]
Statistical Analysis 4: Comparison: Community-based Exercise Group vs Wait-listed Usual Medical Care; Test type: Superiority; p = 0.491, Mixed Models Analysis; Contrasts from a linear mixed models analysis at 6 months adjusted for randomization factors (age, gender, BMI, WOMAC-PF, knee flexion); Mean Difference (Final Values) = -0.8, 98.3% CI 2-sided [-3.7 to 2.0]
Statistical Analysis 5: Comparison: Clinic-based Outpatient Exercise Group vs Community-based Exercise Group; Test type: Superiority; p = 0.021, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.2, 98.3% CI 2-sided [-4.5 to 0.1]
Statistical Analysis 6: Comparison: Clinic-based Outpatient Exercise Group vs Community-based Exercise Group; Test type: Superiority; p = 0.179, Mixed Models Analysis; [statistical method as in outcome 1, analysis 4]; Mean Difference (Final Values) = -1.3, 98.3% CI 2-sided [-3.6 to 1.0]

2. Secondary Outcome: Composite Score of Performed-based Tests of Physical Function.
Description: Scores on 6 performance-based tests (i.e., the 6-minute walk test, 40-meter gait speed, stair ascend/descend test, single leg stance balance test, chair stand test, and floor sitting-rising) were combined into a composite score formed with the unit-weighted Z scores of constituent tests to provide a more representative and stable measure of the subjects' underlying functional performance. The unit weights refer to averaging standardized scores (e.g., the scores for each performance-based test are converted to Z-scores before applying equal weights). Higher Z-scores represent better functional performance. The Z-scores for each participant can be interpreted as deviations from the baseline average of the whole group. We considered a change in Z-score of 0.2 as clinically important because it represents approximately 20% of a standard deviation relative to the baseline average of the whole group.
Time Frame: Baseline, 3 and 6 months
Population: Intention-to-treat approach was used among participants with follow-up data.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Clinic-based Outpatient Exercise Group | Community-based Exercise Group | Wait-listed Usual Medical Care
Number analyzed (Participants) | 96 | 96 | 48
Z-score
  Baseline | 0.02 (0.8) | -0.06 (0.8) | -0.11 (0.7)
  3 months: number analyzed (Participants) | 89 | 87 | 44
  3 months | 0.49 (0.7) | 0.3 (0.8) | 0.13 (0.7)
  6 months: number analyzed (Participants) | 83 | 76 | 40
  6 months | 0.5 (0.8) | 0.36 (0.9) | 0.25 (0.7)
Statistical Analysis 1: Comparison: Clinic-based Outpatient Exercise Group vs Wait-listed Usual Medical Care; Test type: Superiority; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.3, 98.3% CI 2-sided [0.1 to 0.4]
Statistical Analysis 2: Comparison: Clinic-based Outpatient Exercise Group vs Wait-listed Usual Medical Care; Test type: Superiority; p = 0.012, Mixed Models Analysis; [statistical method as in outcome 1, analysis 4]; Mean Difference (Final Values) = 0.2, 98.3% CI 2-sided [0.01 to 0.4]
Statistical Analysis 3: Comparison: Community-based Exercise Group vs Wait-listed Usual Medical Care; Test type: Superiority; p = 0.005, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.2, 98.3% CI 2-sided [0.02 to 0.3]
Statistical Analysis 4: Comparison: Community-based Exercise Group vs Wait-listed Usual Medical Care; Test type: Superiority; p = 0.052, Mixed Models Analysis; [statistical method as in outcome 1, analysis 4]; Mean Difference (Final Values) = 0.2, 98.3% CI 2-sided [-0.003 to 0.3]
Statistical Analysis 5: Comparison: Clinic-based Outpatient Exercise Group vs Community-based Exercise Group; Test type: Superiority; p = 0.015, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.2, 98.3% CI 2-sided [0.02 to 0.3]
Statistical Analysis 6: Comparison: Clinic-based Outpatient Exercise Group vs Community-based Exercise Group; Test type: Superiority; p = 0.489, Mixed Models Analysis; [statistical method as in outcome 1, analysis 4]; Mean Difference (Final Values) = 0.02, 98.3% CI 2-sided [-0.003 to 0.3]

3. Other Pre Specified Outcome: Physical Activity Energy Expenditure - Measured by Portable Activity Monitor (SenseWear).
Description: Real-time measure of daily energy expenditure physical activity assessed by portable activity monitor.
Time Frame: Baseline, 3 and 6 months
Population: Intention-to-treat approach was used among participants with follow-up data.
Measure: Mean (Standard Deviation); unit: Kcal/day
Arm/Group | Clinic-based Outpatient Exercise Group | Community-based Exercise Group | Wait-listed Usual Medical Care
Number analyzed (Participants) | 96 | 96 | 48
Kcal/day
  Baseline: number analyzed (Participants) | 96 | 95 | 47
  Baseline | 511 (411) | 541 (419) | 459 (352)
  3 months: number analyzed (Participants) | 85 | 86 | 43
  3 months | 566 (451) | 547 (407) | 525 (411)
  6 months: number analyzed (Participants) | 84 | 79 | 40
  6 months | 538 (403) | 480 (420) | 509 (518)
Statistical Analysis 1: Comparison: Clinic-based Outpatient Exercise Group vs Wait-listed Usual Medical Care; Test type: Superiority; p = 0.943, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4, 95% CI 2-sided [-106 to 114]
Statistical Analysis 2: Comparison: Clinic-based Outpatient Exercise Group vs Wait-listed Usual Medical Care; Test type: Superiority; p = 0.814, Mixed Models Analysis; [statistical method as in outcome 1, analysis 4]; Mean Difference (Final Values) = 15, 95% CI 2-sided [-112 to 142]
Statistical Analysis 3: Comparison: Community-based Exercise Group vs Wait-listed Usual Medical Care; Test type: Superiority; p = 0.787, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -15, 95% CI 2-sided [-125 to 95]
Statistical Analysis 4: Comparison: Community-based Exercise Group vs Wait-listed Usual Medical Care; Test type: Superiority; p = 0.581, Mixed Models Analysis; [statistical method as in outcome 1, analysis 4]; Mean Difference (Final Values) = -36, 95% CI 2-sided [-164 to 92]
Statistical Analysis 5: Comparison: Clinic-based Outpatient Exercise Group vs Community-based Exercise Group; Test type: Superiority; p = 0.676, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 19, 95% CI 2-sided [-71 to 109]
Statistical Analysis 6: Comparison: Clinic-based Outpatient Exercise Group vs Community-based Exercise Group; Test type: Superiority; p = 0.330, Mixed Models Analysis; [statistical method as in outcome 1, analysis 4]; Mean Difference (Final Values) = 51, 95% CI 2-sided [-52 to 154]

ADVERSE EVENTS:
Time Frame: The adverse events were collected during subjects participation in the study (over 6 months).
Description: The study used a standard questionnaire to monitor AEs every 1.5 months.
Arm/Group | Clinic-based Outpatient Exercise Group | Community-based Exercise Group | Wait-listed Usual Medical Care
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/96 | 0/48
Serious Adverse Events (participants affected / at risk) | 5/96 | 4/96 | 5/48
Other Adverse Events (participants affected / at risk) | 39/96 | 42/96 | 22/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinic-based Outpatient Exercise Group (N=96) | Community-based Exercise Group (N=96) | Wait-listed Usual Medical Care (N=48)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Disorders (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Injury, poisoning and procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Surgical and medical procedures (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinic-based Outpatient Exercise Group (N=96) | Community-based Exercise Group (N=96) | Wait-listed Usual Medical Care (N=48)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (18) | 17 (18) | 8 (8)
Back Pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 9 (9) | 5 (5)
Other musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 13 (13) | 13 (13) | 6 (6)
Cataract (Eye disorders) | 1 (1) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-31): https://cdn.clinicaltrials.gov/large-docs/11/NCT02237911/Prot_SAP_000.pdf